CLINICAL TRIAL: NCT00701324
Title: An Open Phase I Single Dose Escalation Study of Two Dosing Schedules of BI 811283 Administered Intravenously Over 24 h Continuous Infusion in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Brief Title: BI 811283 in Various Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 1247.1; 2007-000191-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Arm A (Experimental): BI 811283, 24h infusion d1 and d15 every 4 weeks
  Interventions: Drug: BI 811283
- Arm B (Experimental): BI 811283, 24h infusion d1 every 3 weeks
  Interventions: Drug: BI 811283

INTERVENTIONS:
Drug: BI 811283 — dose escalation BI 811283, Arm B (3 weeks)
  Arms: Arm B
Drug: BI 811283 — dose escalation BI 811283, Arm A (day 1)
  Arms: Arm A
Drug: BI 811283 — dose escalation BI 811283, Arm A (day 15)
  Arms: Arm A

SUMMARY:
The main objective of this trial is to provide safety data in terms of drug-related adverse events (AE) for the recommendation of the dose for further trials in the development of BI 811283.

Secondary objectives are the collection of antitumour efficacy data and the determination of the pharmacokinetic profile of BI 811283.

ELIGIBILITY:
Inclusion criteria:

Patients with confirmed diagnosis of advanced, non-resectable and/or metastatic solid tumours, who have failed conventional treatment or for whom no therapy of proven efficacy exists or who are not amenable to established treatment options Secure central venous access Evaluable tumour deposits Recovery from reversible toxicities of prior anti-cancer therapies Age >= 18 years Life expectancy >= 6 months Written informed consent in accordance with International Conference on Harmonisation (ICH) guideline for Good Clinical Practice (GCP) and local legislation Eastern Cooperative Oncology Group performance score <= 2

Exclusion criteria:

Serious illness, concomitant non-oncological disease (e.g. active infectious disease), or ongoing toxicity of prior therapies considered by the investigator to potentially compromise patients' safety in this trial Pregnancy or breastfeeding Known brain metastases Second malignancy requiring therapy Left ventricular ejection fraction (LVEF) < 50% in echocardiography or clinical congestive heart failure New York Heart Association grade III - IV Myocardial infarction within the last 6 months prior to inclusion or symptomatic coronary artery disease Absolute neutrophil count less than 1500 / mm3 Platelet count less than 100 000 / mm3 Bilirubin greater than 1.5 mg / dl (> 26 mcmol / L, SI unit equivalent) Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal) Serum creatinine greater than 1.5 mg / dl (> 132 mcmol / L, SI unit equivalent) Women and men who are sexually active and unwilling to use a medically acceptable method of contraception Treatment with other investigational drugs or in another clinical trial within the past two weeks before start of therapy or concomitantly with this trial Chemo-, hormone, radio- or immunotherapy within the past two weeks before start of therapy or concomitantly with this trial Patients unable to comply with the protocol Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 3-4 weeks

SECONDARY OUTCOMES:
Safety profile: incidence and intensity of AEs graded according to the common terminology criteria for AEs, incidence of DLT | throughout the study period
Progression free survival (PFS), Objective response, Response duration, Pharmacodynamic analysis, Basic pharmacokinetics | throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Germany (2):
  - 1247.1.49002 Boehringer Ingelheim Investigational Site, Essen
  - 1247.1.49001 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau

REFERENCES:
- [Derived] Mross K, Richly H, Frost A, Scharr D, Nokay B, Graeser R, Lee C, Hilbert J, Goeldner RG, Fietz O, Scheulen ME. A phase I study of BI 811283, an Aurora B kinase inhibitor, in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2016 Aug;78(2):405-17. doi: 10.1007/s00280-016-3095-6. Epub 2016 Jun 27. PMID 27349901